CLINICAL TRIAL: NCT01680926
Title: Protein-rich Meal Replacement Significantly Reduces Weight, HbA1c and Daily Insulin Requirement Long-term in Patients With Type 2 Diabetes Mellitus and >100 U Insulin Per Day
Brief Title: Metabolic Activation With Almased for Type 2 Diabetes Patients
Acronym: Almased100
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: Almased Wellness GmbH (Industry)
Responsible Party: Principal Investigator, Stephan Martin, Principal Investigator, West German Center of Diabetes and Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Almased100
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; insulin; hbA1c; body weight
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Almased (Experimental): During the first week, all three main meals were replaced with 50 g of a protein-rich meal replacement (Almased) (=1100 kcal per day). During weeks 2-4, only two meals were replaced and a protein-rich lunch was allowed. During weeks 5-12, only dinner was replaced.
  Interventions: Dietary Supplement: Almased

INTERVENTIONS:
Dietary Supplement: Almased — During the first week, all three main meals were replaced with 50 g of a protein-rich meal replacement (Almased) (=1100 kcal per day). During weeks 2-4, only two meals were replaced and a protein-rich lunch was allowed. During weeks 5-12, only dinner was replaced.
  Other Names: Almased-Vitalkost

SUMMARY:
Overweight patients with type 2 diabetes are often being treated with an intensified insulin therapy. However, in many cases, even a high insulin dosage (> 100 U per day) does not achieve satisfying metabolic control. A new therapy option is necessary that makes it possible to lower the daily insulin requirement and to improve metabolic control. The aim of this study was to investigate whether a protein-rich meal replacement is suitable to lower the daily insulin requirement and to reduce HbA1c and body weight.

DETAILED DESCRIPTION:
The pilot study included patients with type 2 diabetes (n=22), that injected >100 U insulin daily. During the first week, all three main meals were replaced with 50 g of a protein-rich meal replacement (Almased) (=1100 kcal per day). During weeks 2-4, only two meals were replaced and a protein-rich lunch was allowed. During weeks 5-12, only dinner was replaced. Clinical parameters were determined at the beginning of the study, after 4, 8 and 12 weeks as well as after 1.5 years of follow-up. Wilcoxon signed rank test was used for the intention-to-treat analysis and Mann-Whitney test for subgroup analyses.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes
* BMI > 27 kg/m2
* age 35-75 years
* insulin therapy >100 U insulin per day

Exclusion Criteria:

* contraindication for a calorie reduced diet

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
insulin demand per day | 12 weeks
  daily insulin dosage

SECONDARY OUTCOMES:
HbA1c | 12 weeks
  HbA1c
body weight | 12 weeks
  body weight

CONTACTS AND LOCATIONS:
Overall Officials: Stepahn Martin, MD, Principal Investigator — West German Center of Diabetes and Health
Locations (1):
- West German Center of Diabetes and Health, Düsseldorf, Germany

REFERENCES:
- See also: Homepage WDGZ — http://www.vkkd-kliniken.de/zentreninstitute/gesundheits_und_therapie_centrum/westdeutsches_diabetes_und_gesundheitszentrum_wdgz/